CLINICAL TRIAL: NCT05475184
Title: A Multicenter, Open-label, Single-arm, Phase 2 Study to Evaluate the Efficacy and Safety of JPI-547, a PARP/TNKS Dual Inhibitor in Platinum-resistant, Advanced/Relapsed Ovarian Cancer Subjects Previously Treated With a PARP Inhibitor
Brief Title: A Study to Evaluate the Efficacy and Safety of JPI-547 in Platinum-resistant, Advanced/Relapsed Ovarian Cancer Subjects Previously Treated With a PARP Inhibitor
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JPI-547-201
Record Dates: First submitted 2022-07-13; First posted 2022-07-26 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: This study will be conducted with subjects with HRD-positive, platinum-resistant, advanced/relapsed ovarian cancer with a history of ARP inhibitor treatment using Simon's optimal two-stage design. When the confirmed response is observed in ≥3 out of 18 subjects who are available for tumor assessment in Stage 1, the subjects will proceed with Stage 2. After additional enrollment of 40 subjects who are available for tumor assessment in Stage 2, the assessment will be conducted to identify that the confirmed response is observed in ≥11 out of the final 58 subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JPI-547 (Experimental)
  Interventions: Drug: JPI-547

INTERVENTIONS:
Drug: JPI-547 — Poly-(ADP-ribose) polymerase (PARP) & tankyrase (TNKS) inhibitor.
  * The investigational product (IP) will be administered once daily for 28 days (4 weeks) with 1 cycle.
  * 1 capsule (JPI-547 150 mg) will be administered once daily at the same time (e.g., a fixed time in the morning) in a fasted condition within 2 hours before or after a meal.

SUMMARY:
To evaluate the efficacy and safety of JPI-547, a PARP/TNKS dual inhibitor in Platinum-resistant, advanced/relapsed ovarian cancer subjects previously treated with a PARP inhibitor

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced/metastatic high-grade serous epithelial ovarian, fallopian tube or primary peritoneal cancer*:

  1. who has undergone ≥2 previous chemotherapy regimen;
  2. with confirmed platinum resistance**;
  3. ≥3 month PARP inhibitor treatment history;
  4. confirmed BRCA1/2 mutation *** or HRD ****
* Subjects with at least one measurable lesion in accordance with RECIST v1.1
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Subjects with life expectancy ≥12 weeks
* Patients with adequate hematologic, kidney, and liver functions confirmed using the following criteria (retesting of laboratory tests is allowed once during screening)
* Subjects who voluntarily decided to participate in this study after being fully informed and gave informed consent

Exclusion Criteria:

* Subjects who meet any of the following conditions cannot participate in this study:

  1. Subjects with a history of severe drug hypersensitivity or the hypersensitivity to IP and its ingredients or similar drugs
  2. Subjects with dysphagia
  3. Subjects confirmed with the following medical or surgical/procedural history:
* Primary malignant tumor other than ovarian cancer diagnosed or treated within 24 months prior to baseline (individuals with successfully treated cutaneous basal/squamous cell carcinoma are eligible for enrollment)
* Major surgery requiring general anesthesia or respiratory support within 4 weeks prior to baseline (2 weeks for video-assisted thoracoscopic surgery [VATS] or open-and-closed [ONC] surgery)
* Severe cardiovascular disease (e.g., myocardial infarction and unstable angina) that occurred within 24 weeks prior to baseline
* New York Heart Association Class 3 or 4 heart failure within 24 weeks prior to baseline
* Severe cerebrovascular disease observed within 24 weeks prior to baseline
* Pulmonary thrombosis or deep vein thrombosis within 24 weeks prior to baseline, or bronchial asthma, obstructive pulmonary disease, or other serious, life-threatening lung disease (e.g., acute respiratory distress syndrome and lung failure) considered ineligible for study participation
* Infections requiring treatment, such as systemic antibiotics and antivirals, within 2 weeks prior to baseline, or other uncontrolled ≥Grade 3 active infectious diseases
* Symptomatic interstitial lung disease
* Subjects who showed poor recovery from hematologic toxicity in the past chemotherapy (e.g., ≥grade 3 toxicity for ≥4 weeks)
* Bone marrow or stem cell transplantation with high-dose chemotherapy
* Total gastrectomy or total duodenectomy
* Individuals with a history of myelodysplastic syndrome (MDS) or pretreatment cytogenetic test results indicating a risk of MDS/acute myeloid leukemia (AML) 4) Subjects with the following concurrent conditions:
* Subjects with clinically significant symptoms or uncontrolled central nervous system or brain metastases (except when systemic corticosteroid administration was stopped at least 4 weeks prior to baseline and was stable for ≥4 weeks)
* Subjects who have confirmed clinically significant conditions in the electrocardiogram (ECG) according to the investigator's judgment
* Uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >90 mmHg)
* Bleeding diatheses
* Active hepatitis B or C virus infection (patients with hepatitis may participate if HBV DNA and HCV RNA are below the lower limit of detection established by the study site)
* Known human immunodeficiency virus infection (HIV) positive
* Subjects with neurological and psychiatric disorders severe enough to affect the study results according to the investigator's judgment 5) Subjects who have the following drug treatment history:
* Subjects who have received chemotherapy†, immunotherapy (including biologics), hormone therapy, or therapeutic/palliative radiotherapy‡ within 4 weeks prior to baseline
* Subjects who require continuous (≥4 weeks) treatment of systemic corticosteroids equivalent to prednisone >10 mg/day
* Subjects who were treated with antithrombotic drugs, including antiplatelet agents and anticoagulants, within 2 weeks from baseline or are expected to be treated with them during the study period (however, low molecular weight heparin [LMWH]) treatment is allowed)
* Subjects who require continuous administration of non-steroidal anti-inflammatory drugs (NSAIDs), which have high risk of bleeding 6) Pregnant or lactating women, or women of childbearing potential who do not intend to abstain or use appropriate contraceptive methods* during the study period and up to 3 months after IP administration *Appropriate contraception: 7) Subjects who have taken or undergone another IP or investigation device within 4 weeks prior to baseline 8) subjects who are judged by the investigator as ineligible for study participation

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | From date of study enroll until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 40 months
  To evaluate the objective response rate (ORR) in accordance with the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.

SECONDARY OUTCOMES:
Anti-tumor activity | From date of study enroll until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 40 months
  To evaluate the anti-tumor activity in accordance with RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Gyeonggi-do, South Korea